CLINICAL TRIAL: NCT06279039
Title: Clinical Observation of Exosomes in Patients After Q-switched Laser Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, dai jie, Nanjing First Hospital, Nanjing First Hospital, Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20230116-06
Record Dates: First submitted 2023-04-06; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Exosome; Skin Regeneration; Laser
Keywords: Exosome; Q-switched laser

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- self half face control method (Experimental): One side of the face was treated with exosome liquid dressing twice a day, and the other side was treated without exosome matrix for 2 weeks. The patients were followed up before treatment and 1, 3，7, 14, 28, and 56 days after treatment
  Interventions: Drug: Exosome liquid dressing

INTERVENTIONS:
Drug: Exosome liquid dressing — This study mainly adopted a randomized double-blind self-half face control method. The double-blind method was that the subjects and researchers did not know the experimental group and the control group. 38 sets of matched use sets (left and right, only the manufacturer knew the specific ingredients) were respectively applied to both sides of the cheeks of patients after Q-switched laser. The blind was unblinded after the experiment.
  Other Names: follow

SUMMARY:
the goal of this half-face controlled study is to evaluate the effect of exosome-containing liquid dressings on the recovery of patients after Nd:YAG laser 532 treatment.

DETAILED DESCRIPTION:
The main objective was to collect patients with fleae or seborrheic keratosis after Q-switched laser treatment, and then to use exosomes or matrix on both sides of the face, and finally to evaluate the effect of exosomes on wound healing and prevention of post-inflammatory hyperpigmentation after Nd:YAG laser 532 treatment

ELIGIBILITY:
Inclusion Criteria:

* It meets the diagnostic criteria of seborrheic keratosis or freckle；
* pepole are able to follow the treatment rules of the study and were followed up for 8 weeks；
* informed consent

Exclusion Criteria:

* History of keloids ;
* Pregnancy or lactation;
* Any cosmetics containing growth factor-related ingredients used within 6 months prior to treatment
* Patients with incomplete observation data and incomplete course of treatment were excluded

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Global Aesthetic Improvement Scale score | 1, 3.5, 7, 14, 28, and 56 days
  The treating physician evaluated the patient's improvement, which was divided into four levels: very improved corresponding, substantial improvement, improvement, no change; Corresponding to the best beauty results, significantly improved but not the best, significantly improved, no change
Dermatology Quality of life index | 1, 3.5, 7, 14, 28, and 56 days
  By answering multiple questions, patients self-rated the impact of their current illness on their lives within a week and scored. The answers were graded on four levels, very serious 3, very serious 2, a little 1, and no 0

SECONDARY OUTCOMES:
post-inflammatory hyperpigmentation | 2.4,8 weeks
  At 2, 4 and 8 weeks of follow-up, melanin index was measured by memetreter (memetreter MX18 cuttometer Dual MPA580, EnviroDerm Services (UK) Ltd) at the same follow-up. Objective evaluation of PIH.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Dai, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Jie Dai, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Polla LL, Margolis RJ, Dover JS, Whitaker D, Murphy GF, Jacques SL, Anderson RR. Melanosomes are a primary target of Q-switched ruby laser irradiation in guinea pig skin. J Invest Dermatol. 1987 Sep;89(3):281-6. doi: 10.1111/1523-1747.ep12471397. PMID 3624901
- [Result] Aurangabadkar SJ. Optimizing Q-switched lasers for melasma and acquired dermal melanoses. Indian J Dermatol Venereol Leprol. 2019 Jan-Feb;85(1):10-17. doi: 10.4103/ijdvl.IJDVL_1086_16. PMID 30027914
- [Result] Kilmer SL, Wheeland RG, Goldberg DJ, Anderson RR. Treatment of epidermal pigmented lesions with the frequency-doubled Q-switched Nd:YAG laser. A controlled, single-impact, dose-response, multicenter trial. Arch Dermatol. 1994 Dec;130(12):1515-9. PMID 7986124
- [Result] Zoumalan CI. Topical Agents for Scar Management: Are They Effective? J Drugs Dermatol. 2018 Apr 1;17(4):421-425. PMID 29601619
- [Result] Stadelmann WK, Digenis AG, Tobin GR. Physiology and healing dynamics of chronic cutaneous wounds. Am J Surg. 1998 Aug;176(2A Suppl):26S-38S. doi: 10.1016/s0002-9610(98)00183-4. PMID 9777970
- [Result] Midwood KS, Williams LV, Schwarzbauer JE. Tissue repair and the dynamics of the extracellular matrix. Int J Biochem Cell Biol. 2004 Jun;36(6):1031-7. doi: 10.1016/j.biocel.2003.12.003. PMID 15094118
- [Result] Theoret CL. The pathophysiology of wound repair. Vet Clin North Am Equine Pract. 2005 Apr;21(1):1-13. doi: 10.1016/j.cveq.2004.11.001. PMID 15691596
- [Result] Toyserkani NM, Christensen ML, Sheikh SP, Sorensen JA. Adipose-Derived Stem Cells: New Treatment for Wound Healing? Ann Plast Surg. 2015 Jul;75(1):117-23. doi: 10.1097/SAP.0000000000000083. PMID 24691309
- [Result] Fraser JK, Wulur I, Alfonso Z, Hedrick MH. Fat tissue: an underappreciated source of stem cells for biotechnology. Trends Biotechnol. 2006 Apr;24(4):150-4. doi: 10.1016/j.tibtech.2006.01.010. Epub 2006 Feb 20. PMID 16488036
- [Result] An Y, Lin S, Tan X, Zhu S, Nie F, Zhen Y, Gu L, Zhang C, Wang B, Wei W, Li D, Wu J. Exosomes from adipose-derived stem cells and application to skin wound healing. Cell Prolif. 2021 Mar;54(3):e12993. doi: 10.1111/cpr.12993. Epub 2021 Jan 17. PMID 33458899
- [Result] Kim J, Kim B, Kim S, Lee YI, Kim J, Lee JH. The effect of human umbilical cord blood-derived mesenchymal stem cell media containing serum on recovery after laser treatment: A double-blinded, randomized, split-face controlled study. J Cosmet Dermatol. 2020 Mar;19(3):651-656. doi: 10.1111/jocd.13063. Epub 2019 Jul 22. PMID 31328871